CLINICAL TRIAL: NCT01570517
Title: Evaluation of the DC Devices IASD System in the Treatment of Patients With Heart Failure With Preserved Ejection Fraction
Brief Title: Feasibility Trial of the DC Devices Interatrial Septal Device (IASD) System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corvia Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-01
Record Dates: First submitted 2012-03-21; First posted 2012-04-04 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device implantation (Experimental): Subjects are implanted with the study device.
  Interventions: Device: IASD System

INTERVENTIONS:
Device: IASD System — Implantation of the DC Devices Inc. IASD System

SUMMARY:
The purpose of this study is to evaluate the safety and potential benefits of the interatrial septal defect (IASD) System in patients with heart failure with preserved ejection fraction.

DETAILED DESCRIPTION:
The study was a multi-center, non-randomized feasibility evaluation of the IASD System at three centers in three countries (Denmark, Australia, and Czech Republic). Relevant ethics committee and competent authority approvals were obtained. The study was conducted in accordance with the Declaration of Helsinki. The protocol required the treatment of a minimum of 5 patients, and allowed up to twenty patients to be enrolled.

The primary objective of the trial was to evaluate the safety and potential benefits of the IASD Device System in the treatment of patients with symptomatic heart failure with preserved ejection fraction, despite optimal medical management.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of HFpEF
* Ejection Fraction of at least 45%
* Imaging and hemodynamic evidence of HFpEF
* History of exercise intolerance
* Symptomatic despite optimal medical management
* Signed study specific informed consent

Exclusion Criteria:

* History of thromboembolic events
* Significant structural heart disease or coronary artery disease
* Contraindicated to study required medication
* Right ventricular dysfunction
* History of greater than mild restrictive or obstructive lung disease
* Life expectancy less than one year for non-cardiovascular reasons
* Known or suspected allergy to implant material
* Fertile women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-05; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Device Events | One month

CONTACTS AND LOCATIONS:
Overall Officials: Jan Komtebedde, DVM, Study Chair — DC Devices
Locations (3):
- David Kaye, Melbourne, Australia
- Homolka Hospital, Prague, Czechia
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Result] Sondergaard L, Reddy V, Kaye D, Malek F, Walton A, Mates M, Franzen O, Neuzil P, Ihlemann N, Gustafsson F. Transcatheter treatment of heart failure with preserved or mildly reduced ejection fraction using a novel interatrial implant to lower left atrial pressure. Eur J Heart Fail. 2014 Jul;16(7):796-801. doi: 10.1002/ejhf.111. Epub 2014 Jun 24. PMID 24961390
- [Result] Malek F, Neuzil P, Gustafsson F, Kaye DM, Walton A, Mates M, Sondergaard L, Ihlemann N, Mariani JA, Reddy V. Clinical outcome of transcatheter treatment of heart failure with preserved or mildly reduced ejection fraction using a novel implant. Int J Cardiol. 2015;187:227-8. doi: 10.1016/j.ijcard.2015.03.198. Epub 2015 Mar 18. No abstract available. PMID 25841123